CLINICAL TRIAL: NCT02713932
Title: The Italian Society of Invasive Cardiology Registry on Percutaneous Aortic Valve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, Luca Testa, Consultant Cardiologist, IRCCS Policlinico S. Donato
Other Study IDs: 84/2010/VE
Record Dates: First submitted 2016-02-27; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency; Transcatheter Aortic Valve Replacement
Keywords: Aortic valve stenosis; Aortic valve regurgitation; Transcatheter aortic valve implantation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transcatheter aortic valve implantation
  Interventions: Device: Transcatheter aortic valve implantation

INTERVENTIONS:
Device: Transcatheter aortic valve implantation

SUMMARY:
The Italian Society of Invasive Cardiology Registry on Percutaneous Aortic Valve is a prospective Italian registry including several centers performing TAVI, collecting baseline, procedural and outcome data.

DETAILED DESCRIPTION:
Aortic valve stenosis is the most common degenerative valve disease in the elderly, the prevalence is about 1-2% in the age group> 65 years and 4% in patients aged> 85. The natural history is characterized by a poor prognosis with a survival rate of 62% at 1 year, 32% at 5 years and 18% at 10 years from symptom onset. Predictors of death were age> of 75 years, poor left ventricular ejection fraction, congestive heart failure, chronic obstructive pulmonary disease, severe mitral regurgitation and pulmonary hypertension.

The gold standard therapy, with improved survival, for severe aortic stenosis is the surgical aortic valve replacement with mechanical or biological prosthesis. Cardiac surgery is therapy of choice for patients with severe aortic valve stenosis with left ventricular dysfunction or when symptomatic for lipothymia or syncope, angina pectoris, heart failure.

Criteria for high surgical risk are: left ventricular failure, coronary artery disease, previous cardiac surgery for coronary artery bypass , chronic obstructive pulmonary disease, and/or advanced age and comorbidity , which can be a contraindication to intervention. Frequently cardiac surgery is not performed in elderly patients for the high surgery risk. In the Euro Heart Survey up to 33% of patients with single valve disease, New York Heart Association class III or IV, were not operated for concomitant disease or reduced life expectancy.

The need to provide a therapeutic option for patients considered at high surgery risk, has stimulated the development of prosthetic valve implantable with a percutaneous transcatheter techniques. The percutaneous treatment of valvular aortic stenosis has potential advantages in terms of reduction of hospitalization of elderly patients with high risk of peri-operative mortality and morbidity, as well as avoiding treatment with oral anticoagulants. The experience up to now is very positive, with immediate favorable results in terms of hemodynamic and clinical improvement. Since the procedure is at initial stage of clinical application, it becomes necessary a uniform and standardized data collection to assess the effectiveness of the procedure, the incidence of acute and late complications, and the performance of the biological valve prosthesis.

The investigators propose the establishment of an observational registry of percutaneous aortic valve replacement performed in the Italian Interventional Cardiology Laboratory.

The objectives are:

* Record the clinical criteria used to asses indication for percutaneous aortic valve replacement in different centers
* Record the anatomical and morphological criteria of vascular access and thoraco abdominal aorta, evaluated with noninvasive and invasive diagnostic tests (echocardiography, multislice angiographic computed tomography, aortography) in particular calcification and tortuosity of aorto-iliac-femoral axis, degree of calcifications of the aortic valve and thoracic aortic wall calcifications.
* Record the types of devices used for percutaneous aortic valve replacement
* Observe different way of procedure (type of access, anesthetic protocols, procedural delay, aortic valvuloplasty, and so forth)
* Follow the procedure-related complications and / or of prosthesis implantation.

  * Acute complications:

    * Cerebral ischemia
    * Arrhythmias
    * Pericardial effusion / cardiac tamponade
    * Aortic valve insufficiency
    * Periprosthesis insufficiency
    * Myocardial ischemia
    * Kidney diseases
    * Conversion to cardiac surgery
    * Complications related to arterial vascular access
  * Late complications

    * Residual aortic valve insufficiency
    * Arrhythmias with need of pacemaker
    * Coronary Ischemia
    * Kidney diseases
    * Endocarditis
* Post Procedure hospital stay
* Evaluate the results at 30 days, 6, 12, 18 and 24 months of follow up:

  * echocardiographic mean transvalvular aortic gradient
  * valvular and/or periprosthesis insufficiency
  * left ventricular ejection fraction
  * Evaluate the clinical outcomes at 30 days, 6, 12, 18 and 24 months of follow up

    * New York Heart Association functional class
    * Medical therapy for heart failure
    * Number of hospitalization for heart failure

Information obtained will be analyzed and used to standardize and make more appropriate indications for percutaneous aortic valve replacement to improve and standardize the protocols of procedure, to assess the immediate and long-term effectiveness of the technique, to monitor acute and late complications related and especially to verify the performance of tissue valves in the medium to long term.

The hemodynamics centers wishing to join the register will send a completed form to the steering committee. Once registered they will receive an identification code and pass word for recording data.

Registration of patients that underwent percutaneous aortic valve replacement with prosthetic heart valves with the CE mark, consecutively enrolled during period of 24 months.

Use of paper and electronic case report forms, divided into 4 parts:

I. Personal details, medical history, clinical assessment / Instrumental II. procedure III. Post-procedure hospital stay (24 hours, 48 hours, discharge) IV. Follow up to 30 days, 6 months, 12 months, 18 months, 24 months

The data will be compiled and analyzed on a quarterly basis and discussed with the participating centers with semi-annual meetings

Primary end-points will be:

1. Feasibility of the procedure (functioning of the device, procedural success)
2. Access through the stenotic native aortic valve
3. Effectiveness of the positioning of the valve
4. Removal of the transport system
5. Procedural success will be determined by the efficacy of the valve system with a reduction of the gradient, and no hemodynamically significant valvular regurgitation, as assessed by angiography and color Doppler echocardiography
6. Major intraprocedural adverse events at 30 days, 3, 6, 12, 18 and 24 months

   1. Major arrhythmias
   2. Myocardial infarction,
   3. Cardiac tamponade
   4. Malfunctioning valve
   5. Emergency surgical aortic valve replacement
   6. Emergency aorto-coronary bypass or percutaneous coronary angioplasty
   7. Cardiogenic shock
   8. Infective endocarditis
   9. Stroke or transient ischemic attacks
   10. Aortic dissection
   11. Dissection of the peripheral vessel
   12. Vascular perforation
   13. Acute occlusion of the artery access
   14. Major bleeding
   15. Death
7. New York Heart Association functional class at 30 days, 6, 12, 18 and 24 months
8. Left ventricle ejection fraction measured by echocardiography at 30 days, 6, 12, 18 and 24 months
9. Valve functioning: valve area, residual mean gradient, aortic regurgitation assessed with color Doppler echocardiography at 30 days, 6, 12, 18 and 24 months
10. Incidence of paravalvular regurgitation at 30 days, 6, 12, 18 and 24 months
11. Incidence of infective endocarditis at 30 days, 6, 12, 18 and 24 months
12. Incidence of vascular complications needs surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom transcatheter aortic valve implantation is attempted at participating center.

Exclusion Criteria:

* None except failure to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom transcatheter aortic valve implantation is attempted at participating center.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Major adverse events | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The decision will be made after study completion.

REFERENCES:
- [Derived] Navarese EP, Zhang Z, Kubica J, Andreotti F, Farinaccio A, Bartorelli AL, Bedogni F, Rupji M, Tomai F, Giordano A, Reimers B, Spaccarotella C, Wilczek K, Stepinska J, Witkowski A, Grygier M, Kukulski T, Wanha W, Wojakowski W, Lesiak M, Dudek D, Zembala MO, Berti S; a Joint Effort of the Italian and Polish Cardiac Interventional Societies. Development and Validation of a Practical Model to Identify Patients at Risk of Bleeding After TAVR. JACC Cardiovasc Interv. 2021 Jun 14;14(11):1196-1206. doi: 10.1016/j.jcin.2021.03.024. PMID 34112454
- [Derived] Berti S, Bedogni F, Giordano A, Petronio AS, Iadanza A, Bartorelli AL, Reimers B, Spaccarotella C, Trani C, Attisano T, Marella Cenname A, Sardella G, Bonmassari R, Medda M, Tomai F, Tarantini G, Navarese EP; Italian Society of Interventional Cardiology-GISEdagger. Efficacy and Safety of ProGlide Versus Prostar XL Vascular Closure Devices in Transcatheter Aortic Valve Replacement: The RISPEVA Registry. J Am Heart Assoc. 2020 Nov 3;9(21):e018042. doi: 10.1161/JAHA.120.018042. Epub 2020 Oct 24. PMID 33103545